CLINICAL TRIAL: NCT05673772
Title: A Multicenter, Randomized Controlled Trial of Preoperative Sequential Short-course Radiation Therapy and Oxaliplatin-based Consolidation Chemotherapy for Locally Advanced Rectal Cancer
Brief Title: Preoperative Sequential Short-course Radiation Therapy and FOLFOX for Locally Advanced Rectal Cancer
Acronym: SOLAR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Collaborators: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Gyu-Seog Choi, M.D., Ph.D, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KNUHCRC007
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Neoadjuvant treatment; short-course radiotherapy; Consolidation chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Short-course radiotherapy and 4 cycles of mFOLFOX6 followed by TME. Adjuvant chemotherapy will be given according to the pathological stage (CR~pStageI: 6 cycles of capecitabine or 4 cycles of 5-FU with leucovorin, pStageII-III: 8 cycles of mFOLFOX6)
  Interventions: Radiation: short-course radiotherapy; Drug: mFOLFOX6; Procedure: TME surgery
- Control group (Active Comparator): Conventional chemoradiotherapy followed by TME. Adjuvant chemotherapy will be given according to the pathological stage (CR~pStageI: 6 cycles of capecitabine or 4 cycles of 5-FU with leucovorin, pStageII-III: 8 cycles of mFOLFOX6)
  Interventions: Radiation: Chemoradiotherapy; Procedure: TME surgery

INTERVENTIONS:
Radiation: short-course radiotherapy — 25 Gy in 5 fractions for 5 days
  Arms: Study group
Drug: mFOLFOX6 — Oxaliplatin 85 mg/m2, Levoleucovorin 200mg (or Leucovroin, Leucosodium 400mg)/m2, 5- FU 400 mg/m2, and continuous 5- FU 2,400 mg/m2 for 46 hours
  Arms: Study group
Radiation: Chemoradiotherapy — 45~50.4 Gy/25fr with concurrent use of either capecitabine or 5-FU+leucovorin(or levoleucovorin or leucosodium)
  Arms: Control group
Procedure: TME surgery — TME surgery

SUMMARY:
The treatment protocol proposed in this study is to perform short-term radiation therapy and 4 cycles of FOLFOX chemotherapy for neoadjuvant treatment of locally advanced rectal cancer. Compared to conventional chemoradiation therapy, the preoperative radiotherapy period is shortened, and the cure rate of rectal cancer patients can be improved by early treatment of micrometastasis using systemic chemotherapy. The patients who are assigned to the study group will received the short-course radiotherapy and 4 cycles of FOLFOX and patients in the control will received conventional chemoradiotherapy for preoperative treatment. All patients are recommended to receive total mesorectal excision (TME) after neoadjuvant treatment and adjuvant chemotherapy will be given according to the pathological stage.

ELIGIBILITY:
Inclusion Criteria:

* Asian
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2
* Pathologically confirmed rectal cancer (rectal cancer located 10 cm or low from the anal verge in pelvis MRI)
* Histologic type: adenocarcinoma, mucinous carcinoma, and signet ring cell carcinoma
* Locally advanced rectal cancer with one or more of the following factors based on pelvis MRI: cTanyN1-2, cT3-4N0, or presence of extramural vascular invasion
* MRI findings such as pelvic lymph node metastasis, anal sphincter invasion, and T4b are not included in the exclusion criteria, which cases will be enrolled by the researcher's discretion
* Patients with appropriate organ (bone marrow, kidney, liver) function
* A person who understands the study and willing to provide informed consent

Exclusion Criteria: (one of the following criteria)

* Colon cancer or rectal cancer located more than 10 cm from the anal verge
* Stage I rectal cancer (clinical stage cT1-2N0)
* Clinically or pathologically diagnosed distant metastasis (cTanyNanyM1)
* Familial adenomatous polyposis
* Hereditary nonpolyposis colorectal cancer
* History of chemotherapy or radiotherapy within 6 months
* History of colorectal cancer or other type of malignancy within 5 years (except for cured nonmelanoma skin or in situ cervical cancer)
* Comorbidities that make it difficult to undergo chemotherapy or radiotherapy
* Bone marrow suppression with neutrophil count <2 ×109/L or platelet count <100 ×109/L prior to the first chemotherapy
* Peripheral sensory neuropathy with functional impairment (grade 2 or higher)
* Severe renal dysfunction (GFR ≤30ml/min by Wright or Cockroft formula)
* Severe hepatic dysfunction
* Genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Taking tegafur, gimeracil, and oteracil potassium complex and those within 7 days of discontinuation
* Taking sorivudine or brivudine
* Significant heart disease or myocardial infarction within the last 6 months
* Hereditary diseases or history of coagulopathy
* Central nervous system disorders with disability or mental disorders
* Pregnant or lactating women
* Currently participating in other clinical trials or receiving research medication
* Unhealed wounds, fractures, peptic ulcer, abscesses in the abdominal cavity
* Active gastrointestinal bleeding
* Active infections requiring antibiotics for injection
* Emergency Surgery
* History of hypersensitivity to the drugs in study protocol
* Patients with non-malignant tumor diseases
* Dihydropyrimidine dehydrogenase deficiency
* Not willing to participate

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2028-12-28 (Estimated); Study Completion 2031-12-28 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival | 3 years
  To compare the 3-year disease-free survival between the experimental arm and the control arm

SECONDARY OUTCOMES:
pCR rate | within 30 days after TME
  CR (complete regression), no tumor cells and only fibrotic mass or acellular mucin pools
Toxicity of neoadjuvant radiotherapy and chemotherapy | 6 months
  Neoadjuvant treatment associated toxicity (Common Terminology Criteria for Adverse Events version v5.0)
R0 resection | within 30 days after TME
  Rate of R0 resection of TME
TRG | within 30 days after TME
  Pathological tumor regression grade (TRG) (Dworak/Mandard/AJCC TRG classification)
Surgical complications | within 60 days after TME
  Surgical complications classified according to the Clavien-Dindo classification
Incidence of peripheral neuropathy | 3 years
  Incidence of oxaliplatin-induced peripheral neuopathy
European Organization for Research and Treatment of Cancer Quality of Life C30 | 2 year after surgery
  The EORTC Core Questionnaire (QLQ-C30) includes six clearly distinguishable functioning scales that have been thoroughly tested and validated on an international level and that are available in 110 different language versions
European Organization for Research and Treatment of Cancer Quality of Life CR29 | 2 year after surgery
  The QLQ-CR29 has five functional and 18 symptom scales. It contains four subscales (urinary frequency (UF), blood and mucus in stool (BMS), stool frequency (SF), and body image (BI)) and 19 single items (urinary incontinence, dysuria, abdominal pain, buttock pain, bloating, dry mouth, hair loss, taste, anxiety, weight, flatulence, fecal incontinence, sore skin, embarrassment, stoma care problems, sexual interest (men), impotence, sexual interest (women), and dyspareunia) [11]. Patients are asked to indicate their symptoms during the past week(s). Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.
Low Anterior Resection Syndrome score | 2 year after surgery
  Low anterior resection syndrome (LARS) score ; 0 to 20 (no LARS), 21 to 29 (minor LARS ) and 30 to 42 (Major LARS )
The International Index of Erectile Function-5 score, retrograde ejaculation | 2 year after surgery
  Quality of life IIEF-5, retrograde ejaculation
5-year disease-free survival | 5 years
  To compare the 5-year disease-free survival between the experimental arm and the control arm
3-year overall survival | 3 years
  To compare the 3-year overall survival between the experimental arm and the control arm
5-year overall survival | 5 years
  To compare the 5-year overall survival between the experimental arm and the control arm
Loco-regional recurrence | 5 years
  To compare the 3 year and 5-year loco-regional recurrence between the experimental arm and the control arm
Distant metastasis | 5 years
  To compare the 3 year and 5-year distant metastasis between the experimental arm and the control arm

CONTACTS AND LOCATIONS:
Locations (9):
- South Korea (9):
  - Gyu seog Choi, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hwasun Hospital, Gwangju
  - Catholic University of Korea Incheon St. Mary's Hospital, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - Asan Medical Center, Seoul
  - , Korea University Anam Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul National University Bundang Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] Kang MK, Park SY, Park JS, Kim HJ, Kim JG, Kang BW, Baek JH, Cho SH, Seo AN, Kim DW, Kim J, Baek SJ, Kim JH, Kim JY, Ha GW, Park EJ, Park IJ, Kim CH, Kang H, Choi GS. Preoperative sequential short-course radiation therapy and FOLFOX chemotherapy versus long-course chemoradiotherapy for locally advanced rectal cancer: a multicenter, randomized controlled trial (SOLAR trial). BMC Cancer. 2023 Nov 3;23(1):1059. doi: 10.1186/s12885-023-11363-7. PMID 37923987